CLINICAL TRIAL: NCT03709940
Title: Brain Connectivity in Attention Deficit Hyperactivity Disorder (ADHD): a Biomarker to Predict Treatment Response
Brief Title: Brain Connectivity in Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: BCADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ConnectADHD
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: longitudinal study; magnetic resonance imaging (MRI); brain connectivity; biomarker; treatment response; methylphenidate; stimulant medication
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate

STUDY DESIGN:
Intervention Model Description: 30 participants with Attention Deficit Hyperactivity Disorder (ADHD) undergo behavioural tests and brain scanning twice, once under placebo and once under an acute dose of methylphenidate (MPH). The order of the tablets is inverted for the second half of the sample, thus the last 30 participants undergo behavioural tests and brain scanning twice, once under an acute dose of MPH and once under placebo. All 60 participants are then treated with a long-acting formulation of MPH used routinely at the Adult ADHD Clinic.
Who Masked: Participant
Masking Description: The first part of the study (DAY 1 and DAY 2) is conceived as a single-blind placebo-controlled cross-over experiment. Participants are blind to the order of the tablets (placebo and MPH). After the two scanning sessions, all 60 participants are started on a long-acting formulation of MPH used routinely at the Adult ADHD Clinic (open trial phase).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo, MPH (Experimental): Dose order: placebo, methylphenidate (MPH)
  Participants receive a placebo tablet (ascorbic acid 50 mgs) on DAY 1 and a clinically effective dose of short-acting MPH (20 mgs) on DAY 2.
  Interventions: Drug: MPH
- MPH, Placebo (Experimental): Dose order: methylphenidate (MPH), placebo
  Participants receive a clinically effective dose of short-acting MPH (20 mgs) on DAY 1 and a placebo tablet (ascorbic acid 50 mgs) on DAY 2.
  Interventions: Drug: MPH

INTERVENTIONS:
Drug: MPH — Participants undergo behavioural tests and brain scanning twice, once under placebo and once under an acute dose of MPH, before starting long-term treatment with a long-acting formulation of MPH used routinely at the Adult ADHD Clinic.
  Other Names: Methylphenidate

SUMMARY:
This study investigates whether a relationship exists between pre-treatment brain characteristics and treatment response in adults with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
There is a pressing need in psychiatry to offer more individualised treatments, and to improve outcomes from clinical trials. This 'individualised medicine' approach requires the development of biomarkers of treatment response.

60 adults with ADHD are recruited from the Adult ADHD Clinic at the Maudsley Hospital, London, United Kingdom.

The study is developed over three sessions, two at baseline (DAY 1 and DAY 2) and one after two months of treatment (follow-up).

The first two sessions are conceived as a single-blind non-randomised placebo-controlled cross-over experiment. The first 30 participants enrolled in the study receive a placebo tablet (ascorbic acid 50 mgs) on DAY 1 before the behavioural assessment and magnetic resonance imaging (MRI) scan. The behavioural assessment and the functional MRI measurements are repeated two days after (DAY 2), under a clinically effective dose (20 mgs) of short-acting methylphenidate (MPH).

The order of the tablets is reverted for the remaining 30 participants to balance any potential expectation and practice effect between the two conditions. Placebo and medication are over-encapsulated with the same red opaque capsules by the pharmacy team. Also, the protocol followed during the two sessions is absolutely identical in respect of timing and tests administered in order to keep the participants blind to the drug condition (medication or placebo).

After the scanning sessions, all the participants receive the same prescription of a long-acting formulation of MPH, according to the clinical guidelines adopted by the Maudsley Hospital. Treatment response is evaluated clinically and behaviourally after 2 months of treatment (follow-up). Pre-treatment brain characteristics are tested as potential predictors (biomarkers) of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* males
* aged 18-45 years old
* intelligent quotient (IQ) > 70 (as measured by WASI)
* diagnosis of ADHD confirmed through clinical assessment (Adult ADHD Clinic)
* non-medicated (stimulant medication-naive or not taking stimulant medication for at least 4 weeks)

Exclusion Criteria:

* no other brain disorders other than ADHD
* no condition precluding MRI scanning (e.g., metallic implants, claustrophobia)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Diffusion imaging-based measurements as statistically significant predictors of treatment response (i.e. of participants' performance on adult ADHD rating scale at follow-up as compared to baseline). | In the month 2-3 following the last scan.
  Diffusion based measurements include specific measures of anatomical connectivity of pathways originating in the frontal lobes, such as the fronto-striatal pathways and the superior longitudinal fasciculus. According to previously published criteria, treatment response is defined as a symptomatic improvement of at least 30%, as measured by participants' performance on adult ADHD rating scale at follow-up as compared to baseline.

SECONDARY OUTCOMES:
Functional connectivity measurements as statistically significant predictors of treatment response (i.e. of participants' performance on adult ADHD rating scale at follow-up as compared to baseline). | In the month 4-5 following the last scan.
  Functional connectivity measurements include the strength of functional connectivity along pathways originating in the frontal lobes, such as the fronto-striatal pathways and the attentive networks. Treatment response is defined as in outcome 1.
Diffusion imaging-based measurements as statistically significant predictors of treatment response defined by a data-driven approach. | In the month 6-7 following the last scan.
  A categorical approach (data-driven analysis using multivariate k-mean clustering) is used to define treatment response on the basis of clinical and behavioural characteristics at follow-up. Clinical characteristics include participants' performance on adult ADHD rating scale at follow-up as compared to baseline, whereas behavioural characteristics include participants' performance on the Qb test at follow-up as compared to baseline.
Functional connectivity measurements as statistically significant predictors of treatment response as defined by a data-driven approach. | In the month 8-9 following the last scan.
  Treatment response is defined as in outcome 3.

CONTACTS AND LOCATIONS:
Overall Officials: Declan Murphy, MD, PhD, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkkinen S, Radua J, Andrews DS, Murphy D, Dell'Acqua F, Parlatini V. Cerebellar network alterations in adult attention-deficit/hyperactivity disorder. J Psychiatry Neurosci. 2024 Jul 3;49(4):E233-E241. doi: 10.1503/jpn.230146. Print 2024 Jul-Aug. PMID 38960626